CLINICAL TRIAL: NCT01377454
Title: Wearable Sensor to Detect Postural Instability in People After Mild Traumatic Brain Injury (mTBI)
Brief Title: Balance and Mild Traumatic Brain Injury (TBI)
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Laurie King, Assistant Professor of Neurology, Oregon Health and Science University
Other Study IDs: 7419
Record Dates: First submitted 2011-06-17; First posted 2011-06-21 (Estimated); Last update posted 2012-08-08 (Estimated); Status verified 2012-08

CONDITIONS: Brain Concussion; Traumatic Brain Injury
Keywords: mTBI; concussion; mild Traumatic Brain Injury; balance; sensors
MeSH Terms: conditions — Brain Concussion; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this pilot project is to determine whether using one inertial sensor on the waist during routine clinical balance testing (i.e. Balance Error Scoring System (BESS)), will be a more immediate, objective, reliable and sensitive way to measure and quantify balance deficits in individuals with mild Traumatic Brain Injury (mTBI).

DETAILED DESCRIPTION:
The purpose of this pilot project is to gather preliminary data to determine whether using one inertial sensor at the waist during the BESS could provide the examiner with a more immediate, objective, reliable and sensitive way to quantify deficits in postural control in the post-concussive population. The investigators hypothesize that the metrics obtained from the iSWAY will be better able to distinguish mTBI subjects from control subjects than the standard clinical assessment. The specific aims are:

1. To determine test-retest and inter-rater reliability of the clinical BESS compared to the instrumented BESS test.
2. To determine if an instrumented BESS can distinguish mTBI from age-matched control subjects better than the commonly used BESS and to determine the best metrics of sway to separate groups.

ELIGIBILITY:
Inclusion Criteria:

* Have a mild Traumatic Brain Injury or Concussion
* Between the ages 12-40 years

Exclusion Criteria:

* Out of age range

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Healthy controls or individuals with mild Traumatic Brain Injury (mTBI) or concussion.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2011-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

REFERENCES:
- [Derived] King LA, Horak FB, Mancini M, Pierce D, Priest KC, Chesnutt J, Sullivan P, Chapman JC. Instrumenting the balance error scoring system for use with patients reporting persistent balance problems after mild traumatic brain injury. Arch Phys Med Rehabil. 2014 Feb;95(2):353-9. doi: 10.1016/j.apmr.2013.10.015. Epub 2013 Nov 5. PMID 24200875